CLINICAL TRIAL: NCT01135121
Title: Pilot Study on the Role of Diaphragm Fatigue in Weaning From Mechanical Ventilation
Brief Title: Role of Diaphragm Fatigue in Weaning From Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Nijmegen (Other)
Responsible Party: Principal Investigator, Leo Heunks, MD PhD, University Medical Center Nijmegen
Other Study IDs: Wean1
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Weaning; Respiratory Muscle Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Weaning failure
- Weaning succes

SUMMARY:
The purpose of this study is to determine whether the diaphragm develops contractile fatigue during a weaning trial and if this is associated with weaning failure.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 year
* mechanical ventilation for at least 3 days
* the treating physician judges the patient to be ready to be weaned from the ventilator
* informed consent

Exclusion Criteria:

* pre-existent muscle disease (congenital or acquired) or diseases / disorders know to be associated with myopathy including auto-immune diseases.
* upper airway / esophageal pathology (i.e. recent surgery, esophageal varices, diaphragmatic hernia)
* recent (< 1 month) nasal bleeding
* phrenic nerve lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients weaning from mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Fatiguability of the diaphragm | Multiple measurements within 24 hours after start of weaning trial

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands